CLINICAL TRIAL: NCT03107806
Title: COMGAMI Continuous Monitoring of Glucose in Acute Myocardial Infarction
Brief Title: Monitoring Glucose Levels in Patients With Myocardial Infarction
Acronym: COMGAMI
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Blood withdrawal problems despite use of different catheters.
Sponsor: Lars Ryden (Other)
Collaborators: Karolinska Institutet (Other); Swedish Heart Lung Foundation (Other)
Responsible Party: Sponsor-Investigator, Lars Ryden, Senior professor, Karolinska Institutet
Organization: Karolinska Institutet (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2011/1446-31/1
Record Dates: First submitted 2013-04-16; First posted 2017-04-11 (Actual); Last update posted 2019-08-15 (Actual); Status verified 2017-04

CONDITIONS: Acute Coronary Syndromes; Hyperglycemia; Hypoglycemia
Keywords: acute coronary syndromes; hyperglycemia; hypoglycemia; continuous glucose monitoring
MeSH Terms: conditions — Acute Coronary Syndrome; Hyperglycemia; Hypoglycemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Glucose monitoring by OptiScanner® (Other): Glucose monitoring and intervention guided by OptiScanner®
  Interventions: Device: OptiScanner®
- Blinded continuous glucose monitoring (Other): Blinded continuous glucose monitoring by OptiScanner® and glucose lowering intervention guided by routine glucose measurements
  Interventions: Device: OptiScanner®

INTERVENTIONS:
Device: OptiScanner® — 1. Glucose monitoring by OptiScanner® for 48 h
  2. Glucose lowering intervention (insulin) guided by OptiScanner®

SUMMARY:
To evaluate the OptiScanner® for continuous glucose monitoring as a tool to optimize glucose levels in patients hospitalized for acute coronary syndromes

DETAILED DESCRIPTION:
Methodology Part a) Explorative Part b) Randomised, parallel-group design

ELIGIBILITY:
Inclusion Criteria:

* Acute coronary syndrome according to the joint recommendations by the European Society of Cardiology (48, 49)
* Signed written informed consent consistent with Helsinki declaration and local legislations prior to participation in the trial.

Exclusion Criteria:

* <18 years old.
* Congestive heart failure.
* Patients who, in the opinion of the investigator, will have difficulties to comply with the protocol (examples: alcohol or drug abuse, psychiatric disorder).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Accuracy of glucose values derived by the new equipment vs. standard lab recordings | During the first part of the study, up to 6 months
  The above specified part of the study is ongoing. Preliminary data confirms accuracy of recorded glucose values but there is a problem with venous access over the intended time of 48 hours. A new type of venous access will be tested and ethics approval has just been accomplished.

SECONDARY OUTCOMES:
Glucose variability | Hospitalization, through study completion, an average of 1 year
  Glucose variability
Number of episodes of Hypoglycemia | Hospitalization, through study completion, an average of 1 year
  No of episodes of hypoglycaemia defined as glucose <3.0 mmol/L with or without symptoms.
Number of episodes of Hyperglycemia | Hospitalization, through study completion, an average of 1 year
  No of episodes of hyperglycemia >12 mmol/L
Work load in nursing staff | Hospitalization, through study completion, an average of 1 year
  Work load in nursing staff, questionnaire
Time in targeted glucose values | Next step after the completion of the first and ongoing part. through study completion, an average of 1 year
  Targets for plasma glucose are defined and the personnel will have support of the new equipment allowing continuous monitoring of glucose levels when adjusting glucose lowering therapy. This will be compared to monitoring with standard, intermittent glucose measuring.

CONTACTS AND LOCATIONS:
Overall Officials: Camilla Hage, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska University hospital, Stockholm, Sweden